CLINICAL TRIAL: NCT04264377
Title: Towards Targeting the ORigin of the Inflammatory Cascade in Allergic Asthma: Cross-talk Between Airway Epithelium and Immune Cells
Brief Title: Towards Targeting the ORigin of the Inflammatory Cascade in Allergic Asthma
Acronym: ORIENT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, Dr. M. van den Berge, University Medical Center Groningen
Other Study IDs: 201900308
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Asthma; Allergic Asthma
Keywords: Epigenetics; Airway wall remodeling
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: 26 healthy subjects
  Interventions: Procedure: Bronchoscopy
- Asthma: 26 subjects with asthma
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy for retrieval of airway cells

SUMMARY:
Allergic asthma is a complex and heterogeneous disease caused by excessive responses to inhaled allergens. Current medication, including corticosteroids and bronchodilators, does not act on the origin of inflammation but rather combats symptoms, leaving many patients uncontrolled. Airway epithelium is critical for the initiation and progression of asthma pathology.

We will include a 52 subjects divided over two groups: ongoing asthma (26 patients) and non-asthmatic healthy controls (26 subjects) in a cross-sectional study. All subjects will be extensively clinically characterized including respiratory symptoms/questionnaires, in- and expiratory CT-scans, and parameters of large and small airway function and inflammation. In addition, blood and nasal epithelial brushes will be obtained to study the genetic and epigenetic mechanisms of asthma. Finally, bronchoscopy with bronchial biopsies and brushes will be performed under conscious sedation. Bronchial biopsies from both patient groups will be used for single cell transcriptional analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

* Age between 18 and 45 years old.
* Smoking history ≤2 packyears.

Specific inclusion criteria for the two groups:

* Group 1. Patients with ongoing asthma

  * Age of onset of asthmatic symptoms: 0 - 18 years.
  * Documented history of asthma diagnosed according to latest GINA guidelines, i.e. respiratory symptoms and either bronchodilator reversibility (improvement in FEV1 of more than 12% of baseline (and at least 200 mL) after inhalation of 800 µg salbutamol).
  * Use of inhaled corticosteroids or either persistent symptoms of wheeze, cough, or dyspnea or regular use of β2 agonists at least once a week during the last 2 months.
  * PC20 methacholine < 8 mg/ml.
* Group 2. Non-asthmatic controls

  * No history of asthma.
  * No use of inhaled corticosteroids or β2-agonists for a period longer than 1 month.
  * No symptoms of wheeze, nocturnal dyspnea, or bronchial hyperresponsiveness.
  * PC20 methacholine > 8 mg/ml, FEV1/FVC > 70% and FEV1 > 80% predicted.

Exclusion Criteria:

* FEV1 <1.2 L,
* Subjects must be able to adhere to the study visit schedule and other protocol requirements.
* A subject is not eligible to enter and participate if he has not signed and dated a written informed consent form prior to participation in the study.
* A subjects is not eligible to enter and participate if he does not agree that we inform his general practitioner.
* Upper respiratory tract infection (e.g. colds), within 6 weeks.
* Serious acute infections (such as hepatitis, pneumonia or pyelonephritis) in the previous 3 months.
* Signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease.
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
* Known recent substance abuse (drug or alcohol).
* Females of childbearing potential without an efficient contraception unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40 mIU/mL or the use of one or more of the following acceptable methods of contraception:

  1. Surgical sterilization (e.g. bilateral tubal ligation, hysterectomy).
  2. Hormonal contraception (implantable, patch, oral, injectable).
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/suppository.
  4. Continuous abstinence.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asthma and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Single-cell transcriptomics bronchial epithelial cell (BEC) | december 2022

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided